CLINICAL TRIAL: NCT04463654
Title: Zero Self-Harm - a Mobile Phone Application to Reduce Non-suicidal Self-injury: A Randomized Clinical Superiority Trial
Brief Title: Zero Self-Harm - a Mobile Phone Application to Reduce Non-suicidal Self-injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 213+983
Record Dates: First submitted 2020-07-07; First posted 2020-07-09 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Self-Injurious Behavior
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zero Self-Harm (Experimental): When randomized to the Zero Self-Harm app the participants will receive an introduction to the app through videos in the app, which explains, amongst others, how to review previous crisis situations and possible strategies for future crisis. This will ensure the navigation and knowledge of the technicalities of the app, in addition to ensure the app can be used privately without personal guidance from e.g a therapist.
  Interventions: Device: Zero Self-Harm app
- Treatment as usual (No Intervention): The control group will continue their present course of treatment and/or counseling at non-profit organizations, service centers in the municipalities, at outpatient treatment services for psychiatric disorders and/or care, attention at emergency departments. They will receive no treatment on the nature of NSSI. Participants in the control group will be offered a possibility to download the Zero Self-Harm app after they have completed the last questionnaire at six months, which will be stressed at the initial appointment as well as after collection of all data.

INTERVENTIONS:
Device: Zero Self-Harm app — Safety plan app for smartphones
  Arms: Zero Self-Harm

SUMMARY:
Non-suicidal self-injury (NSSI), the deliberate, self-inflicted destruction of body tissue without suicidal intent and for purposes not socially sanctioned, is an increasing health care problem in Denmark. Approximately 20 % of Danish adolescents report a history of NSSI at some point in their lives. Individuals with NSSI have an increased risk of suicidality. Therefore, it is of great importance to develop and investigate the effectiveness of a low-cost app in reducing NSSI.

The purpose is to investigate whether treatment as usual (TAU) and the Zero Self-Harm app is superior to TAU in reducing 1) frequency of NSSI-episodes and 2) suicide ideation, and depressive symptoms in individuals with NSSI. As people with NSSI, without a comorbid psychiatric diagnosis, are not eligible to receive psychiatric treatment in Denmark, TAU includes many different treatments and counseling services, i.e. counseling at non-profit organizations, service centers in the municipalities, outpatient treatment services for psychiatric disorders, and care, information and attention at emergency departments. Common to them all is that they do not offer specialized treatment focused on NSSI.

The trial is designed as a 2-arm, parallel group, 6 months, randomized clinical superiority trial. A total of 280 participants, 140 in each arm, will be included. One group will receive TAU, the other will receive TAU and the Zero Self-Harm App. Participants will be recruited through non-profit organizations, service centers in the municipalities, outpatient treatment services, and psychiatric and somatic emergency departments in Denmark.

Inclusion criteria are engagement in two or more episodes of NSSI in the past month, no further planned treatment, have a smartphone, fluent in Danish, provide an informed written consent, age above 18 years.

DETAILED DESCRIPTION:
The purpose of the trial is to investigate whether the introduction of the Zero Self-harm app to individuals with NSSI in Denmark, can 1) reduce the frequency of NSSI-episodes, 2) prevent escalation of NSSI and 3) reduce suicide ideation, and depressive symptoms, compared to treatment as usual.

Hypothesis: The hypothesis is that Zero Self-Harm will reduce the frequency of NSSI-episodes by enhancing participants skills to avoid impulsive urges resulting in NSSI. Thereby, the app will help deal with negative affect and trait impulsivity, core features in the etiology of NSSI, and further decrease associated symptoms, e.g. suicide ideation and depression. We expect that the Zero Self-Harm app will be able to reduce the mean monthly frequency of NSSI in the intervention group by at least 3 episodes. Thus, we hypothesize that the Zero Self-Harm app will be superior to the control condition in 1) reducing the frequency of NSSI-episodes, 2) preventing escalation of NSSI and 3) reducing suicide ideation, and depressive symptoms, compared to treatment as usual.

Methods and design: The trial is designed as a 2-arm, parallel-group, multicentre, pragmatic, randomized clinical superiority trial. Based on the power calculation listed below, a total of 280 participants, 140 in each arm, should be included. One group will receive the Zero Self-Harm app by downloading a specific link sent to them after randomization, and the control group will be allocated to a wait-list and allowed to download the app after they have finished the last questionnaire at 6 months.

Recruitment: Recruitment will be broad and target both individuals with shorter duration and milder symptoms of NSSI, possibly not in contact with mental health facilities, and individuals with more severe and chronic NSSI, already in contact with mental health facilities in Denmark. Recruitment will be done through non-profit organizations, service centres in municipalities, schools for adolescents above 18, outpatient clinics for psychiatric disorders, and psychiatric and somatic emergency departments in Denmark. Recruitment will be conducted through non-profit organizations' websites and social media platforms, as well as providing information about the project through presentations at schools, posters at relevant recruitment facilities and encouraging personnel to refer potential participants when meeting people with NSSI.

Enrolment and randomization: Enrolment will be done by the research assistant when contacted by potential participants via email or telephone. Participants will be encouraged not to send personal information through email and only over the phone, to ensure confidentiality. Potential participants will be given oral and written information about the study, time for consideration and the possibility for an appointment with a next of kin before deciding to enrol in the project. Consent will be obtained by sending an e-mail from REDCap to the trusted Danish secure platform e-boks.

After filling out the baseline questionnaire, participants will be randomly assigned to either the waitlist control group or the Zero Self-harm app, with a 1:1 allocation, using a computer-generated sequence randomization generator in REDCap. The randomization will be stratified by sex and number of previous NSSI-episodes (based on the baseline score of the DSHI) to avoid overrepresentation of patients with a high number og NSSI in one treatment group.

Blinding: Due to the nature of the intervention, neither participants nor the research assistant can be blinded in this trial, and neither primary nor explorative outcomes can be blinded. An employee outside the research team will extract data from REDCap at study completion to two separate excel-sheets, and group allocation will be coded with A and B, to ensure blinding of the research assistant while analysing data, drawing conclusions and drafting the first manuscript. Blinding will be lifted once drafting of the first manuscript has been done.

Intervention: When randomized to the Zero Self-Harm app the participants will receive an email with a link to download the app and an introduction via an instruction manual, in addition to instruction videos implemented in the app. This will ensure the navigation and knowledge of the technicalities of the app. Participants in the waitlist control group will receive no study intervention but will be offered the possibility to download the Zero Self-Harm app after they have finished the last questionnaire at 6 months. This will be stressed at the initial appointment as well as after the collection of data.

Data management: Above-mentioned outcome measures are collected at baseline and 3- and 6-month follow-up through self-administered internet-based questionnaires from REDCap. Participants will receive an e-mail with a link to the online survey, where they can log on to a secure data portal, REDCap, with a personal trial id-number and a two step-code. To improve the response rate, two email reminders are sent out automatically, and if participants still have not answered the questionnaire, they will receive a phone call from the research assistant encouraging them to answer the questionnaire. When data collection is finished, all data from the participants will be imported to a local secured drive with limited access.

Further, there will be a continuous data collection with information about the usage of the app, and register-based data will be collected through the Danish National Hospital Register and the Cause of Death Register. App use and register-based outcomes, such as mortality and admission to psychiatric and/or somatic emergency departments, will be assessed at 3 and 6 months.

To be aware of potential harms of the app, the 20 first participants receiving the Zero Self-harm app will receive a call after they have completed the last questionnaire at 6-months, and interviewed about their experiences of the app. These interviews will be analysed for possible harms, and the results will be discussed in the research group which will then decide on whether or not to continue the trial.

Power analysis: Primary outcome is the mean difference in the monthly frequency of NSSI after 6 months. We expect that participants in the intervention group will have a mean score that is 3.5 points lower compared to participants in the TAU group at follow-up after 6 months. The mean score is based on clinical experience and estimates from a previous study investigating the interventions ability to reduce monthly NSSI episodes (45). Based on previous publications, we expect a post-intervention standard deviation of 9. If the true difference in the experimental and control means is 3.5, we will need to include 140 participants for each group to a total of 280 participants to be able to reject the null hypothesis, that the population means of the experimental and control groups are equal with a probability of 0,1. The Type I error probability associated with this test is 0.05.

Statistical analysis: Analysis of the primary outcome will be conducted according to the intention-to-treat principle: All participants will be included in the final analysis according to group assignment regardless of adherence to treatment. This study has multiple assessment points and for the primary analysis, we will use repeated measurements in a mixed model with unstructured variance. This procedure can handle baseline differences and missing data. For participants with missing data in two or more data points, we will identify potential differences to participants with full data and include these variables as potential confounders in secondary analysis .

Statistical analysis will be conducted in SPSS, version 22.0. Confidence intervals will be presented as well as significance level. All tests will be two-tailed and p values below 0.5 will be considered significant and interpreted with respect to hierarchy of hypothesis recognizing that all outcomes, apart from the primary, are exploratory .

ELIGIBILITY:
Inclusion Criteria:

* Engagement in two or more episodes of NSSI in the past month.
* No further planned treatment focused on NSSI.
* Have a smartphone (IPhone or Android phone).
* Fluent in Danish.
* Skills sufficient to enable use of the Zero Self-Harm app.
* Provide an informed written consent.
* Age ≥ 18 years.

Exclusion Criteria:

* Lack of informed consent.
* Forced care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Deliberate Self Harm Inventory | 6 month
  17-item self-report questionnaire that assesses various aspects of self harm (defined as the deliberate, direct self-destruction of body tissue without suicidal intent) over specified time periods, including frequency (continuous range) and type of self-harm behavior (e.g. cutting, burning etc.). The DSHI demonstrates adequate test-retest reliability and construct, discriminant validity among non-clinical and patient samples

OTHER OUTCOMES:
Becks Suicide Ideation Scale | 6 month
  Becks Suicide Ideation Scale is a 21-item self-report questionnaire measuring suicidal thinking. The outcome is considered as a proxy measure for suicide attempt.
Major Depression Inventory (MDI) | 6 month
  The Major Depression Inventory is a short questionnaire consisting of 12 items capturing depressive symptoms. It can be scored as a diagnostic tool, but also according to severity by a simple sum of the item scores. The minimum score is 0 which indicates no depression and the maximum value is 65 which indicates severe depression.
WHO Well-being Index | 6 month
  The WHO Well-being Index (WHO-5), a widely used short questionnaire to measure quality of life, consisting of 5 simple and non-invasive questions. It is among the most widely used questionnaires assessing subjective psychological well-being.
Rosenberg's Self-Esteem scale | 6 month
  The Rosenberg's Self-Esteem scale consists of 10 items and is a Likert scale. The scale ranges from 0-30. Scores between 15 and 25 are within normal range; scores below 15 suggest low self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Merete Nordentoft, MD, Ph.D MSc, Study Chair — Mental Health Center Copenhagen
Locations (1):
- Kate Trein Andreasson Aamund, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerrero E, Andreasson K, Larsen L, Buus N, Skovgaard Larsen JL, Krogh J, Thastum R, Lindberg L, Lindblad K, Erlangsen A, Nordentoft M. Zero Self-Harm app: a mobile phone application to reduce non-suicidal self-injury-study protocol for a randomized controlled trial. Trials. 2024 Feb 10;25(1):116. doi: 10.1186/s13063-024-07932-1. PMID 38341590